CLINICAL TRIAL: NCT02322307
Title: A Pragmatic Randomized Controlled Trial to Evaluate the Impact of HealthPROMISE Platform on Quality of Care and Quality of Life in Patients With Inflammatory Bowel Disease
Brief Title: Trial on Impact of HealthPROMISE Mobile App on Inflammatory Bowel Disease Care and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GCO 12-1195; 12-0303(1001) (Other: GCO)
Record Dates: First submitted 2014-12-17; First posted 2014-12-23 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis
Keywords: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis; Colitis; PRO; Patient-centric; HealthPROMISE
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Colitis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HealthPROMISE users (Experimental): These are patients who will receive HealthPROMISE application. Patients will be asked to track their quality of life and quality of care using standardized metrics. A combination of different questionnaires (i.e. Short IBD Questionnaire), symptom updates, and IBD quality indicators will be the collected during this study through the HealthPROMISE application.
  Interventions: Other: HealthPROMISE users
- Control Group (Placebo Comparator): After entering baseline questionnaire, control patients get a link to download education application along with PIN. Once patients install app on their devices and use the PIN, the patient is considered to be enrolled in the trial from intention to treat perspective. This control app allows access to patient education content only. There is not any direct feedback on Quality of Life, quality of care and resource utilization.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: HealthPROMISE users — Patients using HealthPROMISE will be asked to use the application once every two weeks at a minimum to provide updates on health information. Providers can use the data entered by patients in real time. Patients will get alerts requesting them to contact their providers if their quality of life scores fall below a certain threshold or their symptoms scores are worrisome. Both patients and physicians are also sent regular notifications with data about their own health or health of their patient panel respectively. Both patients and providers are encouraged to use existing communication tools (phone, office visits, personal health records) since direct patient-physician messaging is not provided in the HealthPROMISE platform. Reminders through app, email and SMS will be used to facilitate patient engagement.
  Physicians will also be encouraged to check the physician panel to see how patients are doing through weekly updates and monthly quality improvement meetings.
  Other Names: HealthPROMISE
  Arms: HealthPROMISE users
Other: Control Group — In order to eliminate a placebo effect, patients in both groups will get an app customized for IBD. Physician and rest of care team will not be blinded since they will use HealthPROMISE dashboard to get alerts and notifications.
  Other Names: InformHealth
  Arms: Control Group

SUMMARY:
HealthPROMISE is a mobile application (app) for patients that allows regular tracking of symptoms by patients and communicates them to physicians. The purpose of this randomized controlled trial is to determine the impact of the HealthPROMISE application on improving patient outcomes. The trial will look at how much patients use the application, whether physicians change treatment in response to new information from patients, and how the patients quality of life change over the span of the study. The investigators hypothesize that HealthPROMISE will enhance physician-patient communication and improve clinical outcomes.

DETAILED DESCRIPTION:
This study will prospectively enroll about 300 patients with Crohn's Disease or Ulcerative Colitis presenting at the Mount Sinai Health System.

Eligible participants who complete the informed consent will fill a Tablet or Web-based questionnaire at the end of which they will be given a pin and offered to download the HealthPROMISE app or an education app. Patients who download HealthPROMISE app will then be requested to provide updates on quality metrics, a quality of life questionnaire, and emergency visits and hospitalizations.

Data will be collected continuously throughout the study using the mobile health app. Study endpoints will primarily be assessed using "intention to treat" analysis. Additionally, per protocol analysis of data will be performed for patients who have logged into the application at least 4 times in 12 months. The total study duration will be 2 years (104 weeks). At 1 year (52 weeks), an interim analysis will be done to determine if study needs to be continued for full 104 weeks. Furthermore, patients in either arm who login using PIN but not completing week 52 (or week 104) exit survey will be considered as "lost to follow up".

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years,
* Internet or Smartphone access
* Ability to complete a Tablet or web-based questionnaire in English language.

Exclusion Criteria:

* Presence of short bowel syndrome, stoma or pouch.
* Presence of a condition or disease that, in the opinion of the investigators, may make it exceedingly difficult for the patient to use HealthPROMISE App, including, but not limited to, advanced dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2015-02; Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Improvement in Quality Indicators (adapted from the American Gastroenterological Association (AGA) outpatient IBD quality metrics and other consensus recommendations) | up to 2 years
  Quality metrics for primary end-point will be adapted from the American Gastroenterological Association (AGA) outpatient IBD quality metrics and other consensus recommendations.

SECONDARY OUTCOMES:
Short Inflammatory Bowel Disease Questionnaire (SIBDQ) | up to 2 years
  The Short Inflammatory Bowel Disease Questionnaire (SIBDQ) is a health-related quality of life (HRQoL) tool measuring physical, social, and emotional status (score 10-70, poor to good HRQoL).
Emergency visits and hospitalizations | up to 2 years
  Number of IBD related emergency visits and hospitalizations
Change in generic QOL score (EQ5D) | at year 1 and at year 2
  The EuroQol (EQ)-5D questionnaire is a simple, generic instrument used to measure health-related quality of life (HRQOL). In a health profile, respondents describe their current health state in 5 dimensions (EQ-5D descriptive system): mobility, self-care, usual-activities (UA), pain/discomfort (P/D), and anxiety/depression (A/D). Problems in these dimensions are classified as none (score = 1), moderate (score = 2), or extreme (score = 3).
Predictors of HealthPromise app utilization (Utilization will be measured through individual logins and data entry in HealthPROMISE app) | up to 2 years
  Utilization will be measured through individual logins and data entry in HealthPROMISE app.

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Atreja, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Atreja A, Khan S, Rogers JD, Otobo E, Patel NP, Ullman T, Colombel JF, Moore S, Sands BE; HealthPROMISE Consortium Group. Impact of the Mobile HealthPROMISE Platform on the Quality of Care and Quality of Life in Patients With Inflammatory Bowel Disease: Study Protocol of a Pragmatic Randomized Controlled Trial. JMIR Res Protoc. 2015 Feb 18;4(1):e23. doi: 10.2196/resprot.4042. PMID 25693610
- See also: Health Promise: Empowering the Doctor and Patient Relationship — http://www.healthpromise.org